CLINICAL TRIAL: NCT02974062
Title: Immediate Effect of Core Stabilization Exercise on Trunk Proprioception in Healthy Individuals: A Feasibility Study
Brief Title: Immediate Effect of Core Stabilization Exercise on Trunk Proprioception in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peemongkon Wattananon (Other)
Responsible Party: Sponsor-Investigator, Peemongkon Wattananon, Principal investigator, Mahidol University
Organization: Mahidol University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2016/016.2601
Record Dates: First submitted 2016-11-21; First posted 2016-11-28 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Back; Instability
Keywords: Position sense; Lumbar stabilization exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lumbar stabilization exercise (Experimental): Lumbar stabilization exercised is a low-intensity exercise that focuses on motor control of deep abdominal and back muscles, rather than their strength or endurance. There are 3 main levels in this exercise; 1) co-contraction of deep abdominal and back muscles, 2) co-contraction with limb movement (self-perturbation), and 3) co-contraction with functional movement (i.e. walking, running, etc.)
  Interventions: Other: Lumbar stabilization exercise
- Healthy control (No Intervention): No intervention was given to this group of participants. They were asked to rest and wait for 15 minutes, then post-test was performed.

INTERVENTIONS:
Other: Lumbar stabilization exercise — Participants were trained using lumbar stabilization exercise based on their initial lumbar stability level. They were received a 30-minute exercise for 1 session in this study.
  Arms: Lumbar stabilization exercise

SUMMARY:
The purposes of this study were to 1) determine test-retest reliability of an iPhone application measurement and protocol, 2) establish minimal detectable change of an iPhone application measurement and protocol, and 3) determine the immediate effect of core stabilization exercise on trunk proprioception in healthy individuals.

DETAILED DESCRIPTION:
This study used a sample of convenience between the ages of 18 - 40. Sixty healthy participants were recruited by flyers posted in 2 Mahidol university physical therapy clinics in Pinklao and Salaya, as well as word of mouth from participants and friend. Sample size calculation was performed using G*Power software (G*Power version 3.1.9.2, University Kiel, Germany). To our knowledge, no study has investigated the immediate effect of core stabilization exercise on trunk proprioception neither in healthy individuals, nor patients with low back pain. However, based on our clinical experiences, we expected to find an improvement (1-tailed) with a medium effect size (Cohen's d = 0.5); therefore, a total of 60 participants were required at confidence level (α) of .05 and power (1-β) of .80.

Participants who were interested in participation underwent a screening process using inclusion-exclusion criteria checklist and receive brief information regarding the study. If they met all inclusion criteria, the consent process was performed. To ensure they understood the study, they were simply asked regarding the study (i.e. objectives, benefits, etc.) before signing the consent form.

After the participants provided a written informed consent, all participants filled out the information sheet for demographic data. After that, they changed their cloth to lab tank top and shorts to expose only their lower back (L1 to S2). The body landmarks, including lumbar spine (L1) and sacrum (S2) were identified and marked with a skin pen for iPhone placement. Each iPhone was placed in the iPhone pocket with transparent film in order to see the iPhone monitor. The pockets were attached to the participant using a Velcro strap around his/her trunk and pelvis. These body landmark identification and iPhone placement process was performed by male or female investigator based upon participant's gender. Once the participant had completed setting up, the data collection process began.

Participants stood on a drawing paper with feet shoulder width apart. The foot print was drawn using a marker. This foot print was used for post-test positioning. The participants stood in a natural stance with arms down by sides. Participants were instructed to stand up straight and maintain that position for recording lumbar and sacral angles in neutral position. After recording, participants were instructed to perform 2 set of 3 repetitions of standing forward bend as far as they can and then return to upright position. Lumbar and sacral angles at full trunk flexion, as well as lumbar and sacral angles at completion of returning to upright were recorded for each repetitions. Data for each set were used to determine test-retest (intra-trial) reliability of an iPhone application, as well as establish minimal detectable change (intra-trial).

Participants underwent trunk proprioception test (pre-test) process by first performing practice trials. Participants performed trunk flexion at 30°, 45°, and 60° (4 repetitions for each degree) with feedback from investigators using those iPhones attached to lumbar spine and sacrum. This practice trials aimed for participants to get familiar with the testing protocol, as well as minimize the learning effect. After completion of practice trials, participants underwent pre-test data collection by perform 3 repetitions of trunk flexion at randomly selected angles each repetition (30°, 45°, and 60°) without feedback. Investigators recorded all lumbar and sacral angle data. After completion of pre-test data collection, all iPhones were removed and body landmarks were erased.

Each participant was randomized into either control or exercise group. Participants in control group waited for 15 minutes (newspaper and magazines were provided during waiting period), while participants in exercise group underwent the assessment of core stability in order to select an appropriate level of core stabilization exercise. After that, each participants in this group received a 30-minute of core stabilization exercise. Clinically, physical therapists would prescribe a 30-minute core stabilization exercise program for patients with non-specific low back pain. This exercise focuses on motor control rather than strength, endurance, or cardiovascular system.37 It is a low intensity exercise to develop an ability to automatically control co-contraction of deep abdominal and back muscles during functional movement. Therefore, the possibility of experiencing muscle fatigue is minimal. However, the participants were instructed to perform stretching exercise after the data collection was completed, and perform in following days as well.

Once participants in control group had finished 15-minute rest, and participants in exercise group had completed core stabilization exercise, they underwent practice trials and post-test data collection using the same protocol starting with marking all body landmarks. Data from test (first 2 sets of 3 repetitions) and retest (last 2 sets of 3 repetitions) from control group were used to determine test-retest (inter-trial) reliability, as well as derive minimal detectable change (inter-trial) of the protocol. Approximate time of the test protocol was 45 minutes including 15-minute rest period for the control group, whereas 60 minutes including 30-minute core stabilization exercise for the exercise group.

Rating of perceived exertion (RPE) and heart rate were used to monitor each participant throughout the protocol to avoid fatigue. Pre- and post-test data from the control and exercise groups were used to determine the immediate effect of core stabilization exercise.

All Statistical analyses were performed using statistical package for the social science (SPSS) software (IBM SPSS Statistics for Windows, Version 21.0. Armonk, New York, USA). Study objective 1 was to determine test-retest reliability of an iPhone application measurement and protocol. Mean angular displacement data from the iPhone application were used to calculate test-retest reliability by using intraclass correlation coefficient (ICC2,k) with confidence intervals. Significance level was held at .05 for all analysis. Study objective 2 was to establish minimal detectable change (MDC) of measurement. Minimal detectable change is defined as the smallest amount of change that likely reflects true change rather than measurement error from the iPhone application and protocol. Study objective 3 was to determine the immediate effect of a 30-minute core stabilization exercise on trunk proprioception in healthy individuals. Prior to utilization of statistical tests, descriptive statistics were performed and statistical assumptions were tested. Transformation will be performed if the data were not normally distributed. Appropriate statistical tests (parametric vs. non-parametric) were performed to determine the effects of 30-minute core stabilization exercise on trunk proprioception. Significance level was held at .05 for all analyses. Post-hoc power analysis was also performed.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 40
* No episode of back pain for 3 months prior to the participation
* No regular exercise routine that is composed of core stabilization exercise We select the age range between 18 and 40 years because one of the previous study demonstrated that patients with non-specific low back pain who had age below 40 years old were more likely to have clinical lumbar instability and would benefit from core stabilization exercise.15 In addition, patients older than 40 years old are more likely to have a specific low back condition,46 such as degenerative spine, spondylosis, or spinal stenosis, which may interfere with our interpretation of the effect of core stabilization exercise on trunk proprioception.

Exclusion Criteria:

* Clinical signs of systemic disease
* Definitive neurologic signs including weakness or numbness in the lower extremity
* Previous spinal surgery
* Diagnosed osteoporosis, severe spinal stenosis, and/or inflammatory joint disease
* Pregnancy
* Any lower extremity condition that would potentially alter trunk movement
* Vestibular dysfunction
* Extreme psychosocial involvement
* Body mass index (BMI) greater than 30 kg/m2
* Active treatment of another medical illness that would preclude participation in any aspect of the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Lumbar position sense | Change from baseline lumbar position sense after receiving a 30-minute lumbar stabilization exercise
  Absolute repositioning error measured by an iPhone application was used to determine change in lumbar position sense after 1 session (30 minutes) of lumbar stabilization exercise

CONTACTS AND LOCATIONS:
Overall Officials: Peemongkon Wattananon, PhD, Principal Investigator — Faculty of Physical Therapy, Mahidol University
Locations (1):
- Faculty of Physical Therapy, Mahidol University, Salaya, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: Yes
All data will be made available for other researchers after the end of the study.

REFERENCES:
- [Background] Hebert JJ, Koppenhaver SL, Magel JS, Fritz JM. The relationship of transversus abdominis and lumbar multifidus activation and prognostic factors for clinical success with a stabilization exercise program: a cross-sectional study. Arch Phys Med Rehabil. 2010 Jan;91(1):78-85. doi: 10.1016/j.apmr.2009.08.146. PMID 20103400
- [Background] O'Sullivan PB. Lumbar segmental 'instability': clinical presentation and specific stabilizing exercise management. Man Ther. 2000 Feb;5(1):2-12. doi: 10.1054/math.1999.0213. PMID 10688954